CLINICAL TRIAL: NCT05155254
Title: An Open-label, Randomized, Phase 3 Clinical Trial of IO102-IO103 in Combination With Pembrolizumab Versus Pembrolizumab Alone in Patients With Previously Untreated, Unresectable, or Metastatic (Advanced) Melanoma (IO102-IO103-013 / MK3475-D18)
Brief Title: IO102-IO103 in Combination With Pembrolizumab Versus Pembrolizumab Alone in Advanced Melanoma (IOB-013 / KN-D18)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IO Biotech (Industry)
Collaborators: Syneos Health (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IO102-IO103-013 / KEYNOTE-D18; 2021-004594-32 (EudraCT Number)
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Melanoma; Unresectable Melanoma
Keywords: Metastatic melanoma; Unresectable melanoma; Immunotherapy; Progression free survival; IO102-IO103; Pembrolizumab
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomised 1:1 to receive either dual-antigen IO102-IO103 in combination with pembrolizumab versus pembrolizumab alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IO102-IO103 + pembrolizumab (Experimental): IO102-IO103 subcutaneous injections (85µg) every 3 weeks for a maximum 35 cycles (up to 2 years treatment). Additional dose given during the induction period on Day 8 of cycles 1 and 2. Each patient can be treated for a maximum of 37 administrations in total (up to 2 years treatment).
  Pembrolizumab 200 mg intravenously every 3 weeks for a maximum of 35 cycles.
  Interventions: Drug: IO102-IO103; Drug: Pembrolizumab
- pembrolizumab (Active Comparator): Pembrolizumab 200 mg intravenously every 3 weeks for a maximum of 35 cycles (up to 2 years treatment).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: IO102-IO103 — IO102-IO103 comprises IDO peptide antigen (IO102) and PD-L1 peptide antigen (IO103) emulsified with adjuvant (Montanide ISA 51 VG) administered subcutaneously
  Arms: IO102-IO103 + pembrolizumab
Drug: Pembrolizumab — Pembrolizumab administered intravenously

SUMMARY:
Phase 3, multicenter, international, open-label, randomized, 2-arm trial investigating the safety and efficacy of IO102-IO103 in combination with pembrolizumab as first-line treatment for patients with previously untreated unresectable or metastatic (advanced) melanoma.

Patients will be stratified on the basis of the following factors; Disease stage: Stage III (unresectable) and IV M1a-b versus stage IV M1c-d and BRAFV600 mutation status: mutated vs wild type.

All patients will receive pembrolizumab 200 mg intravenously every 3 weeks for a maximum of 35 cycles (up to 2 years treatment). Patients randomized to IO102-IO103 dual-antigen, immunotherapeutic arm will also be given IO102-IO103 Q3W with an additional dose given during the induction period on Day 8 of cycles 1 and 2. IO102 IO103 will thereafter be administered subcutaneous every 3 weeks during the maintenance period. Each patient can be treated for a maximum of 37 administrations in total (up to 2 years of treatment).

The primary objective is to investigate the efficacy of IO102-IO103 in combination with pembrolizumab (compared with pembrolizumab alone) in terms of progression free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage III (unresectable) or stage IV melanoma, as per American Joint Committee on Cancer 8th edition guidelines not amenable to local therapy
2. Patients are treatment naive, that is, no previous systemic anticancer therapy for unresectable or metastatic melanoma. For clarification, the following patients are eligible:

   1. Patients with BRAFV600 mutation-positive melanoma are eligible if treatment naive and without rapidly progressive disease as per investigators assessment. Documented BRAF V600 mutation status must be available from all patients prior to trial entry.
   2. Patients who have received previous adjuvant and/or neoadjuvant therapy with targeted therapy or immune therapy are eligible if administered the last dose at least 6 months before inclusion in this trial (randomization), and if relapse did not occur during active treatment or within 6 months of treatment discontinuation.
3. At least 1 measurable lesion according to response evaluation criteria for solid tumors (RECIST v1.1) and confirmed by IRC.
4. Provision of archival (obtained within 3 months), or newly acquired biopsy tissue not previously irradiated, and blood at screening for biomarker assessments. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

Exclusion Criteria:

1. Patients with known or suspected central nervous system (CNS) metastases or with the CNS as the only site of active disease are excluded with the following exception:

   • Patients with controlled (stable) brain metastases will be allowed to enroll (subject to baseline magnetic resonance imaging (MRI) confirmation). Controlled (stable) brain metastases are defined as those with no radiographic progression for at least 4 weeks after radiation and/or surgical treatment at the time of signed informed consent. Patients must have been off steroids for at least 2 weeks before signed informed consent and have no new or progressive neurological signs and symptoms.
2. Patient has received previous radiotherapy within 2 weeks of start of trial treatment (visit 2). Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
3. Patients with BRAFV600-positive disease who are experiencing rapidly progressing disease and/or have received standard first-line therapy with BRAF and/or MEK inhibitor for unresectable or metastatic disease.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 3.5 years
  PFS defined as the time from randomization to the first documented disease progression ((based on Independent Review Committee in accordance with RECIST v1.1) or death from any cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 2.5 years
  ORR defined as the percentage of patients achieving a confirmed PR or CR. ORR will be determined by an IRC in accordance with RECIST v1.1.
Overall survival (OS) | Approximately 5.5 years
  OS defined as the time from randomisation until death from any cause. months. This will be determined by an IRC in accordance with RECIST v1.1.
Durable Objective response rate (DRR) | Approximately 3.5 years
  DRR is defined as the percentage of patients achieving a PR or CR > 6 months. This will be determined by an IRC in accordance with RECIST v1.1.
Complete response rate (CRR) | Approximately 3.5 years
  Percentage of patients with a visit response of CR, which will be determined by the IRC in accordance with RECIST v1.1.
Duration of response (DoR) | Approximately 3.5 years
  DoR will be measured from the date of first observed objective response until disease progression or death (whichever is earlier) (based on IRC).
Time to response (TTR) | Approximately 3.5 years
  TTR is defined as the time from the date of randomization to the date of first observed PR or CR (based on IRC).
Time to complete response (TTCR) | Approximately 3.5 years
  TTCR is defined as the time from the date of randomization to the date of first observed CR (based on IRC).
Disease control rate (DCR) | Approximately 3.5 years
  DCR is defined as the percentage of patients achieving a PR or CR or SD (based on IRC).
Incidence of e.g. AEs and SAEs (Safety and Tolerability) | Approximately 3.5 years
  Incidence of AEs and SAEs, and treatment related AEs and SAEs. Incidence of AEs causing discontinuation of trial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, MD, Prof, Principal Investigator — Institut for Klinisk Medicin, Herlev-Gentofte Hospital; Denmark
Locations (111):
- United States (4):
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - VCU Massey Cancer Center, Richmond, Virginia
- Australia (8):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Sunshine Coast University Hospital, Birtinya
  - Peter MacCallum Cancer Centre PMCC - East Melbourne, Melbourne
- Belgium (2):
  - Universitair Ziekenhuis Gent UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Nikolaas, Sint-Niklaas
- Czechia (4):
  - FNHK Klinika onkologie a radioterapie, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - FN Ostrava, Ostrava
  - FNKV Department of Dermatology, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Herlev og Gentofte Hospital, Herlev
  - Odense University Hospital, Odense
- France (13):
  - Centre Hospitalier Universitaire de Besançon Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire de Bordeaux Hospital Saint Andre, Bordeaux
  - Hopital Ambroise, Boulogne-Billancourt
  - Centre Georges Francois Leclerc, Dijon
  - Chu Grenoble - Hopital Albert Michallon, La Tronche
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital de La Timone, Marseille
  - CHU de Nice Hpital de lArchet 2, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugene Marquis, Rennes
  - Institut de Cancérologie de L'Ouest, Saint-Herblain
  - Centre Hospitalier de Valence (CHV), Valence
  - Gustave Roussy, Villejuif
- Germany (18):
  - Universitatsklinikum Augsburg Medizincampus Sued, Augsburg
  - Charite Universitaetsmedizin Berlin, Berlin
  - St. Josef Hospital - Ruhr-Universitt Bochum, Bochum
  - University Hospital Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - University Hospital Frankfurt Theodor-Stern-Kai, Frankfurt
  - Universitatsklinik fur Dermatologie und Venerologie der MLU Halle-Wittenberg, Halle
  - Elbe Klinikum Buxtehude, Hamburg
  - Nationales Centrum fr Tumorerkrankungen NCT, Heidelberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Department of Dermatology University of Mainz, Mainz
  - Universitatsmedizin Mannheim Dermatologie, Mannheim
  - Mühlenkreiskliniken AöR, University Hospital Ruhr University Bochum Campus Minden, Minden
  - LMU Muenchen, München
  - Universitaetsklinikum Muenster, Münster
  - Hospital Tubingen, Tübingen
  - Universittsklinikum Wuerzburg, Würzburg
- Hungary (3):
  - Orszagos Onkologiai Intezet, Budapest
  - Bor, -Nemikortani es Onkodermatologiai Klinika, Pécs
  - Hetenyi G Korhaz, Onkologiai Kozpont, Szolnok
- Israel (6):
  - Emek Medical Center, Afula
  - Ben-Gurion University of the Negev - Soroka University Medical Center - Soroka Clinical Research Center, Beersheba
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center - The Ella Lemelbaum Institute for Immuno-Oncology, Tel Litwinsky
- Italy (13):
  - Clinica Oncologica, AOU Riuniti ancona, Ancona
  - Centro di Riferimento Oncologico, Aviano
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - IRCCS Ospedale San Raffaele, Candiolo
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Istituto Romagnolo per lo Studio dei Tumori " DINO AMADORI", Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Veneto Oncology Institute, Padua
  - Ospedale S. Maria della Misericordia, Perugia
  - IRCCS Istituti Fisioterapici Ospitalieri, Roma
  - Idi-Irccs, Rome
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
- Netherlands (6):
  - The Netherlands Cancer Institute, Amsterdam
  - AMC Amsterdam, locatie VUMC, Amsterdam
  - LUMC, Leiden
  - UMC Maastricht, Maastricht
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Poland (2):
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Masovian Voivodeship
  - Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu, Poznan
- South Africa (2):
  - Cape Town Oncology Trials (Pty) Ltd., Cape Town
  - Mary Potter Oncology Centre Groenkloof, Pretoria
- Spain (16):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - CH Universitario de A Coruña (CHUAC), A Coruña
  - Hospital Clinic i Provincial, Barcelona
  - Instituto Oncologico Dr. Rosell IOR - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Germans Trias i Pujol HUGTP, ICO-Badalona, Barcelona
  - Hospital Vall d'hebron, Barcelona
  - Hospital General Universitario Gregorio MaraÃ±on, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Clinica Universidad de Navarra, Pamplona
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Miguel Servet University Hospital, Zaragoza
- Turkey (Türkiye) (7):
  - Adana City Education and Research Hospital, Adana
  - Gulhane School of Medicine, Ankara
  - Memorial Ankara Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Ege university Faculty of Medicine, T. Aktas Oncology Hospital, Bornova, Bornova
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
- United Kingdom (3):
  - Guy's Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford